CLINICAL TRIAL: NCT04210310
Title: A Pilot, Proof of Concept, Placebo-controlled, Parallel Study of the Effects of High Dose Intranasal Oxytocin for the Treatment of Tinnitus
Brief Title: High Dose Oxytocin Nasal Spray for Treatment of Tinnitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI departure from the institution.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01381
Record Dates: First submitted 2019-12-12; First posted 2019-12-24 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- high-dose intranasal oxytocin (Experimental): Subjects will be asked to use one spray in one nostril 4 times daily (9AM, 1PM, 5PM and 9 PM). Subjects will take 4 sprays daily of oxytocin for the entire study.
  Interventions: Drug: Oxytocin
- Nasal spray (Placebo Comparator): Subjects swill be asked to use one spray in one nostril 4 times daily (9AM, 1PM, 5PM and 9 PM). The spray can be taken with or without food. Subjects will take 4 sprays daily of the placebo for the entire study.
  Interventions: Other: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin — The investigational product, oxytocin nasal spray (45 units/0.1mL for 38mL) is composed of: oxytocin powder (0.3080g), magnesium chloride crystals (2.3100g), citric acid anhydrous gran. (0.1080g), sodium citrate powder (2.1500g), sterile water for irrigation (38.000mL), and Pcca Mucolox liquid base (3.8000mL). Subjects will be asked to self-administer the study medication with 1 puff in one nostril 4 times per day
  Other Names: Pitocin
  Arms: high-dose intranasal oxytocin
Other: Placebo nasal spray — A placebo nasal spray, consisting of magnesium, chloride crystals, citric acid anhydrous gran., sodium citrate powder, sterile water for irrigation, and Pcca Mucolox liquid base. Both active drug and the placebo will appear identical in the glass bottles. The placebo will be administered in the same manner as the active study drug, with 1 puff in one nostril four times per day.
  Arms: Nasal spray

SUMMARY:
The purpose of this study is to evaluate the effects of high-dose intranasal oxytocin for treating tinnitus. The hypothesis is that high dose intranasal oxytocin can significantly reduce tinnitus severity and disability.

DETAILED DESCRIPTION:
This is a pilot, proof of concept, placebo-controlled, parallel study. Participants will be recruited from NYU Langone Medical Center's Ear, Nose & Throat (ENT) Department and will receive either high-dose intranasal oxytocin or a nasal spray containing Pcca Mucolox and distilled water, serving as the placebo. Long term treatment with high-dose oxytocin (45 IU four times daily) may reduce the frequency and severity of tinnitus, the burden tinnitus symptoms cause patients, and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with continuous perception of subjective tinnitus for ≥ 6 months duration.
* Subjects must have had a normal otolaryngologic evaluation within the past year with no evidence of otitis media or externa, a Tinnitus Handicap Inventory (THI) of > 16.
* Subjects must have tinnitus loudness rating of >4/10.

Exclusion Criteria:

* Subjects who are being treated for tinnitus < 6 months due to the acute nature of their condition
* Subjects who have a slight handicap according to the Tinnitus Handicap Inventory Severity Scale.
* Those with tinnitus of a muscular or vascular etiology
* Subjects with conductive hearing loss, history of migraine, or prior use of oxytocin nasal spray.
* Women of childbearing age will not be approached for participation due to the risk of oxytocin-induced uterine contractions.
* Subjects who suffer from migraines.
* Subjects who have history of pulmonary edema, Congestive Heart Failure, and severe renal disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Newman, MD, Principal Investigator — NYU Langone
Locations (1):
- 222 East 41st Street Ambulatory Care Center, Preston Robert Tisch Center for Men's Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Lawrence.newman@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Period: Overall Study
Arm/Group | High-dose Intranasal Oxytocin | Nasal Spray
Started | 32 | 1
Completed | 0 | 0
Not Completed | 32 | 1
Not completed — Lost to Follow-up | 32 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Intranasal Oxytocin | Nasal Spray | Total
Number analyzed (Participants) | 32 | 1 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.5) | 66 (0) | 60.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 27 | 1 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 1 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale (VAS)-Rated Tinnitus Loudness
Description: Participants use a VAS to rate the loudness of tinnitus on an 11-point Likert scale. Total scores range from 0 (minimum) to 10 (maximum); higher scores indicate greater tinnitus loudness.
  No response to nasal spray is defined as a decrease in VAS Score of less than 2, while a patient-reported improvement is defined as a decrease in VAS Score of more than 3.
Time Frame: Baseline, Week 9
Population: Study was terminated prematurely due to PI and study team departing the institution. Data were not collected for the primary outcome measure.
Arm/Group | High-dose Intranasal Oxytocin | Nasal Spray
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Weeks
Description: Every other week, participants will receive a phone call from study staff to discuss their experience using the study drug and monitor for any adverse effects.
Arm/Group | High-dose Intranasal Oxytocin | Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/1
Other Adverse Events (participants affected / at risk) | 6/32 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Intranasal Oxytocin (N=32) | Nasal Spray (N=1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Intranasal Oxytocin (N=32) | Nasal Spray (N=1)
Mild Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atypical, intermittent chest pain (Cardiac disorders) | 1 | 0
Mild Headache (Nervous system disorders) | 1 | 0
Intermittent Dizziness (Nervous system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Increased urination (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to PI/Study Team departure from institution. No outcome measure data collected or analyzed. All participants lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04210310/Prot_SAP_000.pdf